CLINICAL TRIAL: NCT05619887
Title: Effect of Muscle Reflex Inhibition on Cardiorespiratory Responses to Exercise in Hypoxia
Brief Title: Muscle Reflex Inhibition in Hypoxic Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Phil Ainslie, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Muscle_reflex_hypoxia
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Dyspnea; Muscle Strain
Keywords: Dyspnea; Exercise; Muscle reflex; Type III/IV afferents
MeSH Terms: conditions — Dyspnea; Sprains and Strains; Motor Activity | interventions — Fentanyl; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will complete all interventions (control and experimental) following drug washout.
Who Masked: Participant, Investigator
Masking Description: The participant will not know whether they are receiving placebo or fentanyl. The primary investigator will also no know if the participant is receiving placebo or fentanyl.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Sea level control (Placebo Comparator): Sea level exercise will be completed after the administration of 1 mL of isotonic saline into the intrathecal (spinal) space between L3-L4.
  Interventions: Other: Saline
- Sea level experimental (muscle reflex suppression) (Experimental): Sea level exercise will be completed after the administration of 0.25 mL of fentanyl into the intrathecal (spinal) space between L3-L4.
  Interventions: Drug: Fentanyl
- High altitude control (Placebo Comparator): High altitude exercise will be completed after the administration of 1 mL of isotonic saline into the intrathecal (spinal) space between L3-L4.
  Interventions: Other: Saline
- High altitude experimental (muscle reflex suppression) (Experimental): High altitude exercise will be completed after the administration of 0.25 mL of fentanyl into the intrathecal (spinal) space between L3-L4.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — Fentanyl, when administered into the intrathecal (spinal) space suppresses feedback from the muscles below the site of action, i.e., the legs. It does not affect resting cardiorespiratory responses. We are using this to test what role the muscle reflex plays during exercise.
  Other Names: fentaNYL Citrate
  Arms: High altitude experimental (muscle reflex suppression); Sea level experimental (muscle reflex suppression)
Other: Saline — An equal volume (as above) of saline will be administered into the intrathecal (spinal) space. This has no effect of cardiorespiratory responses at rest or during exercise; it is to control for the invasiveness of the procedure required to suppress muscle feedback in the experimental condition.
  Arms: High altitude control; Sea level control

SUMMARY:
The goal of this interventional study is to compare muscle reflex function under settings of normoxia (normal oxygen level), acute hypoxia (brief oxygen-lack) and chronic hypoxia (long-duration exposure to oxygen-lack).

The main question is: Does the muscle reflex adapt to chronic hypoxia?

Young, healthy participants will complete light-to-high intensity cycling exercise with and without suppression of the muscle reflex. Suppression of the muscle reflex will be via spinal administration of the opioid Fentanyl. In the control condition, saline will be administered into the spinal space. Participants will complete control (saline) and experimental (Fentanyl) exercise conditions at sea-level (Kelowna, BC, Canada) breathing room air and whilst breathing a lower fraction of oxygen (acute hypoxia). Thereafter, participants will complete the exercise test after living at high altitude (White Mountain, CA, USA) for 2 weeks whilst breathing room air (chronic hypoxia) and breathing a higher fraction of oxygen (restored normoxia).

DETAILED DESCRIPTION:
Purpose:

To determine whether muscle reflex control of cardiorespiratory function is sensitized by chronic exposure to low oxygen environments. To do this, fentanyl will be administered into the lumbar spine to suppress nerve activity coming from the muscle during upright cycling exercise.

Hypothesis:

Cardiorespiratory responses (ventilation, blood pressure and heart rate) to cycling exercise will be suppressed when muscle reflex activity is partially blocked with fentanyl administration. This suppression will be augmented in a dose-dependent manner with the duration of hypoxic exposure.

Design:

This is a repeated measures cross-over design with participants completing control (saline) and experimental (fentanyl) conditions both low and high altitude; a total of six visits is required. Sea level testing sessions will involve a cycling exercise bout while breathing room air and a second exercise bout breathing a hypoxic gas mixture meant to simulate the altitude at White Mountain. High altitude testing sessions will involve the same cycling exercise bout while breathing room air and another exercise bout while breathing a hyperoxic gas mixture meant to simulate the altitude in Kelowna. Cardiorespiratory (ventilation, blood pressure and heart rate) will be measured throughout with (fentanyl) and without (saline) muscle reflex suppression. A 7-km time trial test will be performed during each visit to determine how the muscle reflex influences exercise performance.

Experimental procedures:

Participants will visit the lab on six occasions; 3 in both Kelowna and White Mountain. Participants will be requested to practice regular exercise and dietary habits that can be easily replicated in the 24 hours prior to every laboratory visit. Exercise and dietary patterns will be documented during the first visit and thereafter the participants will be reminded of these practices and instructed to match them as closely as possible in the 24 hours leading up to all subsequent visits. Participants will only be instructed to avoid heavy exercise in the 12 hours prior to testing sessions. On the first visit (Kelowna), participants will be introduced into the lab, where we will give oral and written instruction detailing the procedures and associated risks related to participating. Details of the experimental visits are outlined below:

Sea level:

* Familiarization and fitness test (1 h) General introduction to the lab, testing equipment and measurements devices. Maximal aerobic power test on an upright cycle ergometer.
* Main experimental visit #1, saline or fentanyl (2 h) Invasive cannulas will be inserted and drugs administered by an anesthetist. Complete four steady-state exercise bouts (3 min each) while breathing room air.

After a 2 min wash-in, complete four steady-state exercise bouts (3 min each) while breathing hypoxic gas (FiO2 = 0.15).

Complete a 7 km time trial test. - Main Experimental visit #2, Intrathecal (spinal) saline or fentanyl (2 h) Complete identical procedures as experimental visit #1, but the opposite condition.

High altitude:

* High altitude fitness test #1 (30 min) Maximal aerobic power test on upright cycle ergometer.
* Main experimental visit #3, saline or fentanyl (2 h) Invasive cannulas will be inserted and drugs administered by an anesthetist. Complete four steady-state exercise bouts (3 min each) while breathing room air.

After a 2 min wash-in, complete four steady-state exercise bouts (3 min each) while breathing hyperoxic gas (FiO2 = 0.30).

Complete a 7 km time trial test.

- Main experimental visit #4, saline or fentanyl (2 h) Complete identical procedures as experimental visit #3, but the opposite condition.

ELIGIBILITY:
Inclusion Criteria:

* aged 19 - 40 years old
* not taking medications (exception oral contraception)
* no history of cardiovascular, respiratory or neurological disease
* members of the high altitude expedition to White Mountain in 2023

Exclusion Criteria:

* post-menopausal or pregnant
* obese
* current smokers
* taking prescription medications that may affect responses to exercise

All potential participants will be screened by a physician to identify co-morbidities

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Ventilation | Data collected during steady-state breathing in the last minute of exercise
  Ventilation, in liters per minute.

SECONDARY OUTCOMES:
Mean arterial blood pressure (entire pressure wave) | Data collected during steady-state breathing in the last minute of exercise
  Blood pressure, in millimeters of mercury

OTHER OUTCOMES:
Exercise performance | The duration, i.e., however long it takes to complete the exercise; this is typically 7-14 minutes
  Time, in seconds, to complete 7 kilometers of cycling, i.e. a time-trial

CONTACTS AND LOCATIONS:
Overall Officials: Philip N Ainslie, PhD, Principal Investigator — University of British Columbia- Okanagan
Locations (1):
- University of British Columbia - Okanagan Campus, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
No personal data will be made available publicly or to other researchers.

REFERENCES:
- [Result] Amann M, Proctor LT, Sebranek JJ, Pegelow DF, Dempsey JA. Opioid-mediated muscle afferents inhibit central motor drive and limit peripheral muscle fatigue development in humans. J Physiol. 2009 Jan 15;587(1):271-83. doi: 10.1113/jphysiol.2008.163303. Epub 2008 Nov 17. PMID 19015193
- [Result] Wan HY, Weavil JC, Thurston TS, Georgescu VP, Bledsoe AD, Jessop JE, Buys MJ, Richardson RS, Amann M. The muscle reflex and chemoreflex interaction: ventilatory implications for the exercising human. J Appl Physiol (1985). 2020 Oct 1;129(4):691-700. doi: 10.1152/japplphysiol.00449.2020. Epub 2020 Aug 20. PMID 32816637